CLINICAL TRIAL: NCT05954806
Title: Hump-nosed Pit Viper Bite: A Review of Cases to Understand the Clinical Profile of Patients and the Role of Antivenom Administration, at a Tertiary Care Centre in Kerala, South India
Brief Title: Clinical Profile and Antivenom Use in Hump-nosed Pit Viper Bites in Kerala, South India: A Review.
Status: Completed | Type: Observational
Sponsor: Jubilee Mission Medical College and Research Institute (Other)
Responsible Party: Principal Investigator, Siju V Abraham, MD, Associate professor, Jubilee Mission Medical College and Research Institute
Other Study IDs: 87/21/IEC/JMMC&RI
Record Dates: First submitted 2023-06-16; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Envenomation, Snakebite; Envenomation
Keywords: Hump-nosed pit viper; anti venom
MeSH Terms: conditions — Snake Bites

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients With Hypnale Hypnale Bite receiving Antivenom: Patients With Hypnale Hypnale Bite receiving Antivenom for local or systemic signs of envenomation
  Interventions: Drug: Antivenom Snakes
- Patients With Hypnale Hypnale Bite not receiving Antivenom: Patients With Hypnale Hypnale Bite not receiving Antivenom for local or systemic signs of envenomation

INTERVENTIONS:
Drug: Antivenom Snakes — No specific antivenom exists for a bite by Hypnale hypnale yet most patients are treated with non-specific antivenoms, risking reactions without hope of benefit. In this study we compare patients With Hypnale Hypnale Bite receiving Antivenom vrs patients With Hypnale Hypnale Bite not receiving Antivenom.
  Other Names: The polyvalent f(ab')2 antibody
  Groups: Patients With Hypnale Hypnale Bite receiving Antivenom

SUMMARY:
Several controversies exist in Hypnale bite management in Kerala. Even though leading bodies like WHO recommend against using antivenom for hypnale bites, many physicians still administer antivenom for snakebites even when the culprit snake is identified. Anecdotal experience suggests that the reasons for doing so range from lack of confidence in the identification of the snake, confusion as to whether or not to approach it syndromically and symptomatically rather than relying on the species identification, doubts as to whether there exists para-specific neutralization capability for the available polyvalent antivenom and fear of medicolegal culpability in denying antivenom in a case of 'snake envenomation'. To date, these domains and rationale have not been studied. It is also to be kept in mind that the evidence behind the WHO recommendation against the use of antivenom in Hypnale is based on expert opinion and case reports. The investigators intend to compare clinical manifestation and outcome amongst Hypnale hypnale bite patients who received the polyvalent antivenom to those who did not.

The investigators also intend to describe the clinical and laboratorical profile of patients with Hypnale hypnale envenomation .

DETAILED DESCRIPTION:
Hump-nosed pit viper bites are the second most common snakebite presented to our institute as evidenced by the data in our snakebite registers. Acute kidney injury is reported in nearly 10% of the cases in our institute.

Since 2016, the participating institute maintains a snakebite register that records the patient's name, hospital number, date and time of the bite, hospital admission, and snake identification data after expert confirmation, if done. The investigators intend to review the cases with confirmed Hypnale envenomation and describe the clinical and laboratory profile of patients and their course of hospitalization.

Hump-nosed pit viper envenomation, the venom components, and the pharmacodynamics of the venom are unique to the region that it has missed the attention of many experts in the field. The current available polyvalent antivenom does not utilize the venom of Hypnale. Yet, antivenom is used by physicians for snakebites even when the culprit snake is identified, citing many reasons. The reasons range from snake misidentification to doubts as to whether para-specific neutralization capability exists for the available polyvalent antivenom. Often fear of medicolegal culpability in denying antivenom in a case of 'snake envenomation', and confusion as to whether or not to approach it syndromically and symptomatically rather than relying on the species identification also comes into play.

ELIGIBILITY:
- Inclusion Criteria:

Case records of all snakebite in which the specimen brought is identified as Hump-nosed pit viper (Hypnale hypnale)

Exclusion Criteria:

* Incomplete case records from which no meaningful data can be abstracted.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Hypnale hypnale bite that were treated at a tertiary care centre in central Kerala, India during the period from April 2017 to December 2021.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2022-03-12 (Actual); Primary Completion 2022-06-12 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Mortality among patients administered antivenom compared to those who did not received the antivenom | 3 months
  Mortality among patients administered antivenom compared to those who did not received the antivenom for local or systemic signs of envenomation
Morbidity among patients administered antivenom compared to those who did not received the antivenom | 3 months
  Morbidity among patients administered antivenom compared to those who did not received the antivenom for local or systemic signs of envenomation

SECONDARY OUTCOMES:
Clinical profile of patients with Hypnale hypnale envenomation | 3 months
  Clinical profile of patients with confirmed bite Hypnale hypnale with regards to local or systemic signs of envenomation
Laboratorical profile of patients with Hypnale hypnale envenomation | 3 months
  Laboratorical profile of patients with confirmed bite Hypnale hypnale with regards to local or systemic signs of envenomation

CONTACTS AND LOCATIONS:
Overall Officials: Siju V Abraham, MD, Principal Investigator — Jubilee Mission Medical College and Research Institute
Locations (1):
- Jubilee Mission Medical College and Research Institute, Thrissur, Kerala, India